CLINICAL TRIAL: NCT02489669
Title: Renal Insufficiency Following Contrast Media Administration Trial III (REMEDIAL III): Renalguard System Versus Left-ventricular End-diastolic Pressure-guided Hydration in High-risk Patients for Contrast-induced Acute Kidney Injury
Brief Title: Renal Insufficiency Following Contrast Media Administration Trial III
Acronym: REMEDIALIII
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Clinica Mediterranea (Other)
Responsible Party: Principal Investigator, Carlo Briguori, MD, PhD, Clinica Mediterranea
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCT004
Record Dates: First submitted 2015-06-08; First posted 2015-07-03 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Contrast Nephropathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LVEDP-guided group (No Intervention): Patients allocated to the LVEDP-guided group will continue to receive intravenous 0.9% sodium chloride, according to the protocol suggested in the POSEIDON trial (that is, 5 mL/kg/hr for LVEDP ≤12 mmHg; 3 mL/kg/hr for 13-18 mmHg; and 1.5 mL/kg/h for >18 mmHg). The fluid rate will be eventually modified at the start of the procedure in case of discordance between non-invasive and invasive LVEDP pressure estimate, being the invasive value considered as gold-standard. The fluid rate will continued during the procedure, and for 4 hours post-procedure.
- Renalguard group (Experimental): Patients enrolled in this group will be treated by hydration with 0.9% saline controlled by the RenalGuard system. On top of the 1.5-5.0 ml/kg/h that patients would have received over the previous hour (according to the non-invasive estimate LVEDP), an initial bolus of 250 ml will be administered. In case of LV ejection fraction ≤30% and/or LVEDP >18 mm Hg the bolus will 150 mL. Therefore, furosemide (0.25 mg/kg) will be administered in order to achieve the optimal urine flow rate (≥300 mL/h). The controlled hydration by the RenalGuard system will be continued during the procedure and for 4 hours following the procedure. Urine flow rate is monitored and maintained at the target value through the procedure and during the following 4 hours. Additional furosemide doses are allowed in case of decrease of the urine flow rate below the target value.
  Interventions: Device: RenalGuard system™® (PLC Medical Systems, Inc. Franklin, MA, USA)

INTERVENTIONS:
Device: RenalGuard system™® (PLC Medical Systems, Inc. Franklin, MA, USA) — Patients in the RenalGuard group will be treated by hydration with normal saline controlled by the RenalGuard system™® (PLC Medical Systems, Inc. Franklin, MA, USA). The RenalGuard system includes a) a closed loop fluid management system; b) a high volume fluid pump, c) a high accuracy dual weight measuring system; d) motion detection artifact reduction; e) a single use intravenous set and urine collection system that interfaces with a standard Foley catheter; f) real-time display of urine and replacement fluid volume; g) a timely alerts to drain the urine bag or to replace the hydration fluid bag; f) and safety features such as automatic air and occlusion detection.
  Arms: Renalguard group

SUMMARY:
The urine flow rate (UFR)-guided and the left-ventricular end-diastolic pressure (LVEDP)-guided hydration regimens have been proposed to prevent contrast-induced acute kidney injury (CI-AKI). The REnal Insufficiency Following Contrast MEDIA Administration TriaL III (REMEDIAL III) trial is a randomized, multicenter, investigator-sponsored trial aiming to compare these 2 hydration strategies in high risk patients.

Patients with estimated glomerular filtration rate <45 ml/min/1.73 m2 and/or a high risk for CI-AKI (as defined according to both Mehran's score ≥11 and/or Gurm's score >7) will be enrolled. Patients will be divided in high (>12 mm Hg) and normal LVEDP, non-invasively estimated by transmitral flow velocity to annular velocity ratio (E/E' index). Patients in each group will be randomly assigned to 1) LVEDP-guided hydration with normal saline (LVEDP-guided group). The fluid infusion rate will be adjusted according to the LVEDP as follows: 5 mL/kg/hr for LVEDP <12 mmHg; 3 mL/kg/hr for 13-18 mmHg; and 1.5 mL/kg/hr for >18 mmHg. 2) UFR-rate guided hydration (RenalGuard group). In this group, hydration with normal saline plus low-dose of furosemide is controlled by the RenalGuard system, in order to reach and maintain a high (>300 mL/h) UFR. In all cases iobitridol (an low-osmolar, non ionic contrast agent) will be administered. The primary endpoint is the composite of CI-AKI (i.e., serum creatinine increase ≥ 25% and ≥ 0.5 mg/dl from the baseline value at 48 hours after contrast media exposure) and/or acute pulmonary edema.

DETAILED DESCRIPTION:
Contrast-induced acute kidney injury (CI-AKI) is a powerful predictor of unfavorable early and late outcome. Hydration represents the cornerstone in CI-AKI prevention1. However, at present there is no consensus on how hydration should be carried out. The most recommended hydration regimen is normal saline infusion at 1 mL/kg/h 12 hours before and 12 hours after CM exposure. Limitations of this hydration regimen include 1) preclusion in urgent/emergent settings, and 2) suboptimal efficacy in high- and very high risk patients. Indeed, in high and very-high risk patients the rate of CI-AKI may be still high, whereas a forced hydration regimen may increase the risk of pulmonary edema.

In order to clarify how to carry out optimal hydration, 2 regimens have been recently proposed: 1) left ventricular end-diastolic pressure (LVEDP)-guided hydration and 2) urine flow rate (UFR)-guided hydration. The POSEIDON trial demonstrated that the left ventricular end-diastolic pressure (LVEDP)-guided hydration is superior to the conventional hydration regimen in preventing CI-AKI. In the LVEDP-guided hydration, the fluid infusion rate was adjusted according to the LVEDP as follows: 5 mL/kg/hr for LVEDP <12 mmHg; 3 mL/kg/hr for 13-18 mmHg; and 1.5 mL/kg/hr for >18 mmHg. The reported rate of pulmonary edema was 1.5%.

Another theory for CI-AKI prophylaxis suggests to induction and maintenance of a high UFR. This high UFR should allow the body to rapidly eliminate contrast media, reducing contact time within nephron. The RenalGuard™ System (PLC Medical Systems, Inc.) in combination with limited (0.25 mg/kg) dose of furosemide induces an maintains a high UFR (>300 mL/h) safely by maintaining the intravascular blood volume and minimizing the risk of over or under-hydration. Furthermore, the reported rate of pulmonary edema was <1%.

The purpose of the present study is to compare the LVEDP-guided hydration and the UFR-guided hydration in patients at high risk for CI-AKI.

Following enrollment, patients will be randomly assigned to one of the following treatments: 1) LVEDP-guided group, and 2) RenalGuard group. Enrolled patients will be stratified, according to the estimated LVEDP value, into high LVEDP and normal LVEDP group. LVEDP will be non-invasively estimated by the transmitral flow velocity to annular velocity ratio (E/E' index). Estimated LVEDP pressure >12 mm Hg will be considered high. Patients allocated in both groups will receive intravenous 0.9% sodium chloride for at least one hour prior to cardiac catheterization. In both groups the fluid rate will be adjusted according to the non-invasive LVEDP estimate as follows: 5 mL/kg/hr for LVEDP ≤12 mmHg; 3 mL/kg/hr for 13-18 mmHg; and 1.5 mL/kg/h for >18 mmHg, as suggested in the POSEIDON trial. Invasive LVEDP measurement will be also estimated in all patients by placing an angled 5 or 6-French pigtail catheter in the mid-cavity of the left ventricle at the beginning of the procedure and before contrast media injection in order to confirm the non-invasive estimated value.

The sample size was calculated to demonstrate the superiority of the RenalGuard therapy over the LVEDP-guided hydration regimen. The investigators expect a reduction in the primary composite endpoint from 9% in the LVEDP-guided group to 5% in the RenalGuard group. Using a two-sided Chi-square test with a significance level of 0.05, a total of at least 750 randomized patients (350 in each arm) afforded the study 80% power. The endpoints will be analyzed in the global population and also in the subgroups stratified according to the LVEDP value.

Serum creatinine, cystatin C, blood urea nitrogen, sodium and potassium will be measured the day before, 12, 24, 48 hours and 1 week after administration of the contrast agent; additional measurements will be performed in all cases of deterioration of baseline renal function. CI-AKI is defined as an increase of serum creatinine >=0.3 mg/dl at 48 hours after contrast media exposure.

Patient demographic details, medical history, current medication, eGFR, risk score for CI-AKI, and left ventricular ejection fraction are recorded at baseline. Total hydration volume administered according to the prophylaxis and during the 24 and 48 hours following the procedure as well as the total urine volume will be recorded. The pre-procedure sCr level is considered as the sCr concentration before the initiation of any prophylaxis. End-point data and adverse events are collected during the in-hospital stay and at 1-month. Six-month and 12-month MAE will be also collected. All adverse events are recorded in the case report form and the data coordinating center will be informed by facsimile within 72 hours of any events. Serious events and any other safety issues will be reviewed by an independent Data Monitoring and Safety Committee. All events will be adjudicated by a Clinical Events Committee (CEC), who is blinded to treatment assignment. At least 2 members of the CEC review clinical data and relevant documentation and determine whether end points have occurred according to the study definitions. In case of disagreement between reviewers, a third member of the CEC will adjudicate and the data will be considered by the entire committee if 2 of the 3 reviewers do not agree.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with chronic kidney disease (CKD) scheduled for coronary and/or peripheral angiography and/or angioplasty with an eGFR <45 ml/min/1.73 m2 and/or
* At high risk for CI-AKI according to Mehran's score ≥11 and/or Gurm's score >7

Exclusion Criteria:

* Age <18 years
* Women who are pregnant
* Acute pulmonary edema
* Acute myocardial infarction
* Recent contrast media exposure
* End-stage CKD on chronic dialysis
* Multiple myeloma
* Current enrolment in any other study when enrolment in the REMEDIAL III would involve deviation from either protocol
* Cardiogenic shock
* Administration of theophilline, dopamine, mannitol and fenoldopam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2015-07-15 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Composite of 1) development of CI-AKI, and/or acute pulmonary edema. | within 48 hours after contrast media exposure
  The primary outcome measure is composite of 1) development of CI-AKI, and/or acute pulmonary edema. CI-AKI is defined as an increase in the serum creatinine concentration >=25% and >=0.5 mg/dl from the baseline value at 48 hours after administration of the contrast media or the need for dialysis

SECONDARY OUTCOMES:
Creatinine change | 48 hours
  an increase in the serum creatinine concentration >=0.3 mg/dl at 48 hours after contrast exposure
Cystatin C change | 48 hours
  changes in the serum cystatin C concentration at 24 and 48 hours after contrast exposure
Dialysis rate | 5 days
  the rate of acute renal failure requiring dialysis (defined as a decrease in renal function necessitating acute hemodialysis, ultrafiltration or peritoneal dialysis within the first 5 days post-intervention)
Major adverse event rate | 12 months
  the rate of in-hospital, 6 and 12-month major adverse events (MAE), including death, renal failure requiring dialysis, acute pulmonary edema, and sustained kidney injury. Sustained kidney injury is defined as a persistent ≥25% GFR compared to baseline at the last available value during the follow up.
Length of in-hospital stay (LOS) | 30 days
  the length of in-hospital stay (LOS), calculated as the sum of the number of days since admission until discharge from the hospital.
Impact of LVEDP | 48 hours
  the occurrence of the primary endpoint in the 2 groups stratified according to the LVEDP

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Briguori, Principal Investigator — Clinica Mediterranea

REFERENCES:
- [Result] McCullough PA. Contrast-induced acute kidney injury. J Am Coll Cardiol. 2008 Apr 15;51(15):1419-28. doi: 10.1016/j.jacc.2007.12.035. PMID 18402894
- [Result] Tepel M, Aspelin P, Lameire N. Contrast-induced nephropathy: a clinical and evidence-based approach. Circulation. 2006 Apr 11;113(14):1799-806. doi: 10.1161/CIRCULATIONAHA.105.595090. No abstract available. PMID 16606801
- [Result] Briguori C, Visconti G, Rivera NV, Focaccio A, Golia B, Giannone R, Castaldo D, De Micco F, Ricciardelli B, Colombo A. Cystatin C and contrast-induced acute kidney injury. Circulation. 2010 May 18;121(19):2117-22. doi: 10.1161/CIRCULATIONAHA.109.919639. Epub 2010 May 3. PMID 20439784
- [Result] Solomon R, Werner C, Mann D, D'Elia J, Silva P. Effects of saline, mannitol, and furosemide on acute decreases in renal function induced by radiocontrast agents. N Engl J Med. 1994 Nov 24;331(21):1416-20. doi: 10.1056/NEJM199411243312104. PMID 7969280
- [Result] Brar SS, Aharonian V, Mansukhani P, Moore N, Shen AY, Jorgensen M, Dua A, Short L, Kane K. Haemodynamic-guided fluid administration for the prevention of contrast-induced acute kidney injury: the POSEIDON randomised controlled trial. Lancet. 2014 May 24;383(9931):1814-23. doi: 10.1016/S0140-6736(14)60689-9. PMID 24856027
- [Result] Stevens MA, McCullough PA, Tobin KJ, Speck JP, Westveer DC, Guido-Allen DA, Timmis GC, O'Neill WW. A prospective randomized trial of prevention measures in patients at high risk for contrast nephropathy: results of the P.R.I.N.C.E. Study. Prevention of Radiocontrast Induced Nephropathy Clinical Evaluation. J Am Coll Cardiol. 1999 Feb;33(2):403-11. doi: 10.1016/s0735-1097(98)00574-9. PMID 9973020
- [Result] Briguori C, Visconti G, Focaccio A, Airoldi F, Valgimigli M, Sangiorgi GM, Golia B, Ricciardelli B, Condorelli G; REMEDIAL II Investigators. Renal Insufficiency After Contrast Media Administration Trial II (REMEDIAL II): RenalGuard System in high-risk patients for contrast-induced acute kidney injury. Circulation. 2011 Sep 13;124(11):1260-9. doi: 10.1161/CIRCULATIONAHA.111.030759. Epub 2011 Aug 15. PMID 21844075
- [Result] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- [Result] World Medical Association Inc. Declaration of Helsinki. Ethical principles for medical research involving human subjects. J Indian Med Assoc. 2009 Jun;107(6):403-5. No abstract available. PMID 19886379
- [Result] Anello C, O'Neill RT, Dubey S. Multicentre trials: a US regulatory perspective. Stat Methods Med Res. 2005 Jun;14(3):303-18. doi: 10.1191/0962280205sm398oa. PMID 15969305
- [Result] Kasner M, Westermann D, Steendijk P, Gaub R, Wilkenshoff U, Weitmann K, Hoffmann W, Poller W, Schultheiss HP, Pauschinger M, Tschope C. Utility of Doppler echocardiography and tissue Doppler imaging in the estimation of diastolic function in heart failure with normal ejection fraction: a comparative Doppler-conductance catheterization study. Circulation. 2007 Aug 7;116(6):637-47. doi: 10.1161/CIRCULATIONAHA.106.661983. Epub 2007 Jul 23. PMID 17646587
- [Result] Ommen SR, Nishimura RA, Appleton CP, Miller FA, Oh JK, Redfield MM, Tajik AJ. Clinical utility of Doppler echocardiography and tissue Doppler imaging in the estimation of left ventricular filling pressures: A comparative simultaneous Doppler-catheterization study. Circulation. 2000 Oct 10;102(15):1788-94. doi: 10.1161/01.cir.102.15.1788. PMID 11023933
- [Result] How to diagnose diastolic heart failure. European Study Group on Diastolic Heart Failure. Eur Heart J. 1998 Jul;19(7):990-1003. doi: 10.1053/euhj.1998.1057. No abstract available. PMID 9717033
- [Result] Gurm HS, Dixon SR, Smith DE, Share D, Lalonde T, Greenbaum A, Moscucci M; BMC2 (Blue Cross Blue Shield of Michigan Cardiovascular Consortium) Registry. Renal function-based contrast dosing to define safe limits of radiographic contrast media in patients undergoing percutaneous coronary interventions. J Am Coll Cardiol. 2011 Aug 23;58(9):907-14. doi: 10.1016/j.jacc.2011.05.023. PMID 21851878
- [Result] Ware LB, Matthay MA. Clinical practice. Acute pulmonary edema. N Engl J Med. 2005 Dec 29;353(26):2788-96. doi: 10.1056/NEJMcp052699. No abstract available. PMID 16382065
- [Result] Dorval JF, Dixon SR, Zelman RB, Davidson CJ, Rudko R, Resnic FS. Feasibility study of the RenalGuard balanced hydration system: a novel strategy for the prevention of contrast-induced nephropathy in high risk patients. Int J Cardiol. 2013 Jun 20;166(2):482-6. doi: 10.1016/j.ijcard.2011.11.035. Epub 2011 Dec 26. PMID 22204847
- [Result] Marenzi G, Ferrari C, Marana I, Assanelli E, De Metrio M, Teruzzi G, Veglia F, Fabbiocchi F, Montorsi P, Bartorelli AL. Prevention of contrast nephropathy by furosemide with matched hydration: the MYTHOS (Induced Diuresis With Matched Hydration Compared to Standard Hydration for Contrast Induced Nephropathy Prevention) trial. JACC Cardiovasc Interv. 2012 Jan;5(1):90-7. doi: 10.1016/j.jcin.2011.08.017. PMID 22230154
- [Derived] Hashimoto H, Yamada H, Murata M, Watanabe N. Diuretics for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2025 Jan 29;1(1):CD014937. doi: 10.1002/14651858.CD014937.pub2. PMID 39878152